CLINICAL TRIAL: NCT00144794
Title: Mucopolysaccharidosis I (MPS I) Registry
Status: Recruiting | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: DIREGC07008; U1111-1294-8266 (Registry Identifier: ICTRP)
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Mucopolysaccharidosis I (MPS I)
Keywords: Hurler's Syndrome; Hurler-Scheie Syndrome; Scheie Syndrome
MeSH Terms: conditions — Mucopolysaccharidosis I

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The Mucopolysaccharidosis I (MPS I) Registry is an ongoing, observational database that tracks the outcomes of patients with MPS I. The data collected by the MPS I Registry will provide information to better characterize the natural history and progression of MPS I as well as the clinical responses of patients receiving enzyme replacement therapy, such as Aldurazyme (Recombinant Human Alpha-L-Iduronidase), or other treatment modalities.

The objectives of the Registry are:

* To evaluate the long-term effectiveness and safety of Aldurazyme® (laronidase)
* To characterize and describe the MPS I population as a whole, including the variability, progression, and natural history of MPS I
* To help the MPS I medical community with the development of recommendations for monitoring patients and reports on patient outcomes to optimize patient care

DETAILED DESCRIPTION:
The MPS I Registry is an international program; in addition to the central contact information provided under the "Location" heading, patients may contact:

* In Asia-Pacific - Vivian Liu, +65-6431-2548, Vivian.liu@genzyme.com
* In Europe - +31-35-699-1232, europe@mpsiregistry.com
* In Latin America - +617-591-5500, help@mpsiregistry.com
* In North America - +617-591-5500, help@mpsiregistry.com

ELIGIBILITY:
Inclusion Criteria:

* All patients with a confirmed diagnosis of MPS I are eligible for inclusion. Confirmed diagnosis is defined as: A. documented biochemical evidence of a deficiency in alpha (a)-L-iduronidase enzyme activity and/or B. mutation(s) in the gene coding for a-L-iduronidase, or measurable clinical signs and symptoms of MPS I
* For all patients there should be a completed patient authorization form

Exclusion Criteria:

* No exclusion criteria for participation in the MPS I Registry. NOTE: Registry participation does not exclude participation in other clinical studies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Patients with MPS I
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2003-11-20 (Actual); Primary Completion 2034-01-31 (Estimated); Study Completion 2034-01-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the long-term effectiveness of Aldurazyme | Approximately 17 Years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (180):
- United States (66):
  - Phoenix Children's Hospital- Site Number : 840003, Phoenix, Arizona
  - Arkansas Childrens Hospital- Site Number : 840109, Little Rock, Arkansas
  - Southern California Permanente Medical Group- Site Number : 840108, Los Angeles, California
  - USC Health Sciences Center Dept of Genetics- Site Number : 840082, Los Angeles, California
  - Children's Hospital Oakland- Site Number : 840029, Oakland, California
  - Children's Hospital of Orange County- Site Number : 840074, Orange, California
  - Stanford Unviersity MC Dept of Genetics- Site Number : 840022, Palo Alto, California
  - UC Davis MIND Institute- Site Number : 840010, Sacramento, California
  - Loma Linda University Children's Hospital- Site Number : 840117, San Bernardino, California
  - University of California at San Diego- Site Number : 840007, San Diego, California
  - University of California at San Francisco- Site Number : 840051, San Francisco, California
  - Children's Hospital Colorado - Aurora- Site Number : 840069, Aurora, Colorado
  - University of Colorado at Denver Genetics Site Number : 840068, Aurora, Colorado
  - Yale - Site Number : 840047, New Haven, Connecticut
  - Children's National Medical Center- Site Number : 840067, Washington D.C., District of Columbia
  - University of Florida Dept of Genetics- Site Number : 840083, Gainesville, Florida
  - University of Florida Pediatrics Genetics- Site Number : 840121, Jacksonville, Florida
  - The Atwal Clinic- Site Number : 840112, Jacksonville, Florida
  - University Of Miami SOM- Site Number : 840006, Miami, Florida
  - Pediatric Endocrine Associates- Site Number : 840017, Tampa, Florida
  - Emory University School of Medicine- Human Genetics- Site Number : 840060, Decatur, Georgia
  - Ann and Robert Lurie Children's Hospital- Site Number : 840011, Chicago, Illinois
  - Rush University Medical Center Genetics- Site Number : 840079, Chicago, Illinois
  - Indianapolis University School of Medicine- Site Number : 840027, Indianapolis, Indiana
  - University of Iowa- Site Number : 840032, Iowa City, Iowa
  - University of Louisville- Genetics- Site Number : 840030, Louisville, Kentucky
  - Ochsner Medical Center - Site Number : 840120, New Orleans, Louisiana
  - John Hopkins- Site Number : 840044, Baltimore, Maryland
  - Massachusetts General Hospital-Genetics- Site Number : 840062, Boston, Massachusetts
  - Boston Children's Hospital - PIN- Site Number : 840093, Boston, Massachusetts
  - Baystate Health- Site Number : 840002, Springfield, Massachusetts
  - University of Michigan Pediatrics- Site Number : 840107, Ann Arbor, Michigan
  - Children's Hospital of Michigan- Site Number : 840066, Detroit, Michigan
  - Children's Health Care- Site Number : 840114, Minneapolis, Minnesota
  - University of Minnesota Medical Center Pediatrics- Site Number : 840076, Minneapolis, Minnesota
  - Washington University of St. Louis- Site Number : 840100, St Louis, Missouri
  - University of Nebraska Medical Center- Pediatrics- Site Number : 840084, Omaha, Nebraska
  - Children's Specialty Center of Nevada- Site Number : 840008, Las Vegas, Nevada
  - Joseph M. Sanzari Children's Hospital- Site Number : 840101, Hackensack, New Jersey
  - Atlantic Health System- Site Number : 840099, Morristown, New Jersey
  - St. Peter's University Hospital- Site Number : 840016, New Brunswick, New Jersey
  - St. Joseph's Children's Hospital- Site Number : 840057, Paterson, New Jersey
  - Northwell Health- Site Number : 840102, Manhasset, New York
  - New York University School Of Medicine- Site Number : 840040, New York, New York
  - Metropolitan Hospital Center- Site Number : 840110, New York, New York
  - University of Rochester Medical Center SOM- Site Number : 840105, Rochester, New York
  - State University of New York- Site Number : 840052, Syracuse, New York
  - Duke University Medical Center Genetics Dept- Site Number : 840037, Durham, North Carolina
  - Cincinnati Children's Hospital-Genetics- Site Number : 840041, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center- Site Number : 840119, Cleveland, Ohio
  - Nationwide Children's Hospital - PIN- Site Number : 840091, Columbus, Ohio
  - LSD Data Registry Site LLC- Site Number : 840094, Dublin, Ohio
  - Oregon Health & Science University (OHSU)- Site Number : 840080, Portland, Oregon
  - Children's Hospital of Philadelphia HUP Medical Genetics- Site Number : 840089, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia- Site Number : 840034, Philadelphia, Pennsylvania
  - University of Pittsburgh- Site Number : 840023, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Genetics- Site Number : 840053, Providence, Rhode Island
  - Greenwood Genetcs- Site Number : 840055, Greenville, South Carolina
  - Baylor Research Center- Site Number : 840058, Dallas, Texas
  - University of Utah Health Hospital- Site Number : 840092, Salt Lake City, Utah
  - University of Virginia School of Medicine-Pediatrics- Site Number : 840078, Charlottesville, Virginia
  - Children's Hospital of the Kings Daughters- Site Number : 840072, Norfolk, Virginia
  - Seattle Children's Hospital- Site Number : 840028, Seattle, Washington
  - University Of Washington Medical Center- Site Number : 840059, Seattle, Washington
  - Multicare Health System ¿ Mary Bridge Childrens Hospital- Site Number : 840115, Tacoma, Washington
  - Children's Hospital of Wisconsin-Pediatrics- Site Number : 840054, Milwaukee, Wisconsin
- Argentina (2):
  - Investigational Site Number : 153032, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Investigational Site Number : 153130, Buenos Aires
- Australia (2):
  - Investigational Site Number : 151069, Westmead, New South Wales
  - Investigational Site Number : 152096, Brisbane, Queensland
- Belgium (4):
  - Investigational Site Number : 150944, Brussels
  - Investigational Site Number : 150517, Brussels
  - Investigational Site Number : 151668, Leuven
  - Investigational Site Number : 154008, Roeselare
- Brazil (4):
  - Centro de Pesquisa Clínica Prédio 21, 2o andar Hospital de Clínicas de Porto Alegre- Site Number : 076001, Porto Alegre, Rio Grande do Sul
  - Hospital e Maternidade Celso Pierro - PUC-Campinas- Site Number : 076007, Campinas, São Paulo
  - Instituto Fernandes Figueira - FIOCRUZ- Site Number : 076004, Rio de Janeiro
  - Instituto de Genética e Erros Inatos do Metabolismo- Site Number : 076002, São Paulo
- Canada (9):
  - Investigational Site Number : 124014, Calgary, Alberta
  - Investigational Site Number : 124002, Edmonton, Alberta
  - Investigational Site Number : 124011, Vancouver, British Columbia
  - Investigational Site Number : 124019, Winnipeg, Manitoba
  - Investigational Site Number : 124022, Moncton, New Brunswick
  - Investigational Site Number : 124021, London, Ontario
  - Investigational Site Number : 124006, Toronto, Ontario
  - Investigational Site Number : 124018, Montreal, Quebec
  - Investigational Site Number : 124001, Sherbrooke, Quebec
- Chile (2):
  - Investigational Site Number : 152001, Talcahuano, Región del Biobío
  - Investigational Site Number : 152003, Los Ángeles
- Investigational Site Number : 170001, Bogotá, Colombia
- Investigational Site Number : 1910001, Zagreb, Croatia
- Investigational Site Number : 150659, Prague, Czechia
- Investigational Site Number : 151229, København Ø, Denmark
- Egypt (2):
  - Investigational Site Number : 818002, Cairo
  - Investigational Site Number : 818001, Cairo
- France (6):
  - Investigational Site Number : 250004, Bordeaux
  - Investigational Site Number : 250001, Bron
  - Investigational Site Number : 250002, Marseille
  - Investigational Site Number : 250003, Paris
  - Investigational Site Number : 250005, Paris
  - Investigational Site Number : 250006, Vandœuvre-lès-Nancy
- Germany (2):
  - Investigational Site Number : 151368, Hamburg
  - Investigational Site Number : 150031, Mainz
- Investigational Site Number : 344001, Kowloon, Hong Kong
- Investigational Site Number : 3480005, Pécs, Hungary
- India (4):
  - Investigational Site Number : 356003, Ahmedabad
  - Investigational Site Number : 356001, Kolkata
  - Investigational Site Number : 3560004, Secunderabad
  - Investigational Site Number : 356002, Vellore
- Investigational Site Number : 360001, Jakarta, Indonesia
- Investigational Site Number : 154161, Dublin, Ireland
- Italy (9):
  - Investigational Site Number : 380004, Cusano Milanino, Milano
  - Investigational Site Number : 380002, Ancona
  - Investigational Site Number : 380009, Florence
  - Investigational Site Number : 380003, Genova
  - Investigational Site Number : 380007, Milan
  - Investigational Site Number : 380005, Napoli
  - Investigational Site Number : 380008, Padua
  - Investigational Site Number : 380006, Roma
  - Investigational Site Number : 380001, Udine
- Japan (2):
  - Investigational Site Number : 392102, Nangoku-shi, Kochi
  - Investigational Site Number : 392101, Tokyo
- Investigational Site Number : 154225, Kuwait City, Kuwait
- Investigational Site Number : 4220004, Beirut, Lebanon
- Malaysia (2):
  - Investigational Site Number : 458001, Jalan Pahang
  - Investigational Site Number : 458002, Kuala Lumpur
- Netherlands (2):
  - Investigational Site Number : 151171, Amsterdam
  - Investigational Site Number : 152029, Rotterdam
- Pakistan (2):
  - Investigational Site Number : 154264, Lahore
  - Investigational Site Number : 154266, Lahore
- Investigational Site Number : 608001, Manila, Philippines
- Investigational Site Number : 150575, Warsaw, Poland
- Investigational Site Number : 6200002, Coimbra, Portugal
- Investigational Site Number : 154177, Cluj-Napoca, Romania
- Russia (2):
  - Investigational Site Number : 643001, Moscow
  - Investigational Site Number : 643002, Moscow
- Saudi Arabia (2):
  - Investigational Site Number : 682001, Al Qaţīf
  - Investigational Site Number : 682004, Mecca
- Investigational Site Number : 702001, Singapore, Singapore
- Investigational Site Number : 703001, Bratislava, Slovakia
- South Korea (11):
  - Investigational Site Number : 154286, Changwon-si, Gyeongsangnam-do
  - Investigational Site Number : 153178, Yangsan, Gyeongsangnam-do
  - Investigational Site Number : 154148, Yangsan, Gyeongsangnam-do
  - Investigational Site Number : 153180, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 153196, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 153191, Daejeon
  - Investigational Site Number : 153225, Jeonnam
  - Investigational Site Number : 153192, Seoul
  - Investigational Site Number : 151149, Seoul
  - Investigational Site Number : 153212, Seoul
  - Investigational Site Number : 153222, Seoul
- Investigational Site Number : 7520001, Stockholm, Sweden
- Taiwan (13):
  - Investigational Site Number : 154093, Chiayi City
  - Investigational Site Number : 152152, Hualien City
  - Investigational Site Number : 152244, Kaohsiung City
  - Investigational Site Number : 152246, Kaohsiung City
  - Investigational Site Number : 151534, New Taipei City
  - Investigational Site Number : 151500, Putz City, Chia-yi
  - Investigational Site Number : 151181, Taichung
  - Investigational Site Number : 151179, Taichung
  - Investigational Site Number : 153248, Tainan
  - Investigational Site Number : 152153, Tainan
  - Investigational Site Number : 151182, Taipei
  - Investigational Site Number : 152321, Taipei
  - Investigational Site Number : 153158, Taoyuan
- Thailand (5):
  - Investigational Site Number : 764002, Bangkok
  - Investigational Site Number : 764003, Bangkok
  - Investigational Site Number : 764004, Bangkok
  - Investigational Site Number : 764001, Bangkok
  - Investigational Site Number : 764005, Khon Kaen
- United Kingdom (8):
  - Investigational Site Number : 152287, Birmingham, England
  - Investigational Site Number : 151646, London, London, City of
  - Investigational Site Number : 150303, London, London, City of
  - Investigational Site Number : 152361, Salford, Manchester
  - Investigational Site Number : 150455, Manchester, Missouri
  - Investigational Site Number : 154240, Birmingham
  - Investigational Site Number : 152156, Glasgow
  - Investigational Site Number : 151123, London
- Vietnam (2):
  - Investigational Site Number : 154212, Hanoi
  - Investigational Site Number : 704002, Ho Chi Minh City

REFERENCES:
- [Background] Viskochil D, Muenzer J, Guffon N, Garin C, Munoz-Rojas MV, Moy KA, Hutchinson DT. Carpal tunnel syndrome in mucopolysaccharidosis I: a registry-based cohort study. Dev Med Child Neurol. 2017 Dec;59(12):1269-1275. doi: 10.1111/dmcn.13545. Epub 2017 Sep 11. PMID 28892147
- [Background] Arn P, Bruce IA, Wraith JE, Travers H, Fallet S. Airway-related symptoms and surgeries in patients with mucopolysaccharidosis I. Ann Otol Rhinol Laryngol. 2015 Mar;124(3):198-205. doi: 10.1177/0003489414550154. Epub 2014 Sep 11. PMID 25214650
- [Background] Beck M, Arn P, Giugliani R, Muenzer J, Okuyama T, Taylor J, Fallet S. The natural history of MPS I: global perspectives from the MPS I Registry. Genet Med. 2014 Oct;16(10):759-65. doi: 10.1038/gim.2014.25. Epub 2014 Mar 27. PMID 24675674